CLINICAL TRIAL: NCT01610687
Title: A Double Blind, Randomised, Parallel Group, Placebo Controlled Trial of a Combination of THC and CBD in Patients With Multiple Sclerosis, Followed by an Open Label Assessment and Study Extension
Brief Title: A Long-term Safety Extension Study of Delta-9-tetrahydrocannabinol (THC) and Cannabidiol (CBD) in Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWMS0001 EXT
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis; Spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GW-1000-02 (Experimental): Active treatment
  Interventions: Drug: GW-1000-02

INTERVENTIONS:
Drug: GW-1000-02 — Contained THC and CBD as extract of Cannabis sativa L. Each 100 μl actuation delivered a dose containing 2.7 mg THC and 2.5mg CBD. The maximum permitted dose was eight actuations (22 mg THC and 20 mg CBD) in any three hour period, and 48 actuations (130 mg THC and 120 mg CBD) in any 24 hour period.
  Other Names: Sativex

SUMMARY:
An extension study to evaluate the long-term safety, tolerability and efficacy of GW-1000-02 treatment in multiple sclerosis.

DETAILED DESCRIPTION:
Patients who participated in the placebo controlled phase of this study and opted to continue receiving open label GW-1000-02 entered the follow-on extension of the study and completed symptom assessments to determine whether they were continuing to receive clinical benefit from GW-1000-02.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* Multiple Sclerosis of any type.
* Stable Multiple Sclerosis symptomatology during the four weeks before study entry.
* Symptoms of the required severity (>50 mm on a 100 mm Visual Analogue Scale severity scale) in least one of the specified impairment categories; spasticity, muscle spasms, disturbed bladder control, neuropathic pain, limb tremor.
* A stable medication regime during the four weeks before study entry.
* Willing to abstain from cannabis or cannabinoids for at least seven days before study entry, and during the study.
* Agreed either to use effective contraception during the study and for three months thereafter, or had been surgically sterilised or, if female, were post-menopausal.
* Clinically acceptable laboratory results for pre-study screening.
* Willing and able to undertake and comply with all study requirements.
* Willing and able to read, consider and understand the subject information and consent form and give written informed consent. Subjects unable to read or to sign the document procedures were treated as detailed in the Declaration of Helsinki.
* Willing for their general practitioner, and consultant if appropriate, to be informed of study participation.
* Willing for their name to be notified to Home Office for participation in the study.

Exclusion Criteria:

* Known or strongly suspected to be abusing drugs, including alcohol.
* Not prepared to abstain from cannabis or cannabinoids during the study.
* Current or past addiction to cannabis.
* Known or suspected to have had an adverse reaction to cannabinoids causing psychosis or other severe psychiatric illness.
* History of any type of schizophrenia, any other psychotic illness, or other significant psychiatric illness or personality disorder other than depression associated with chronic illness.
* Received any drug containing levodopa (Sinemet®, Sinemet plus®, Levodopa®, L-dopa®, Madopar®, Benserazide®).
* Serious cardiovascular disorder including angina, uncontrolled hypertension, or an uncontrolled symptomatic cardiac arrhythmia.
* Significant renal or hepatic impairment as shown in medical history or indicated by laboratory results.
* History of epilepsy.
* Terminal illness or other condition in which placebo medication would be inappropriate.
* Pregnant, lactating or at risk of pregnancy.
* Participated in any other clinical research study during the 12 weeks before study entry.
* Planned hospital admission between study entry and Visit 6.
* Planned travel outside the UK between study entry and Visit 6.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2001-07; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rivermead Rehabilitation Centre, Oxford, United Kingdom

REFERENCES:
- [Result] Wade DT, Makela PM, House H, Bateman C, Robson P. Long-term use of a cannabis-based medicine in the treatment of spasticity and other symptoms in multiple sclerosis. Mult Scler. 2006 Oct;12(5):639-45. doi: 10.1177/1352458505070618. PMID 17086911

RESULTS

PARTICIPANT FLOW:
Groups:
- GW-1000-02: GW-1000-02 contains Δ tetrahydrocannabinol, 27 mg/ml and cannabidiol, 25 mg/ml as extract of Cannabis sativa L. Subjects received study medication delivered in 100 μl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three hour period and 48 actuations (THC 130 mg:CBD 120 mg) in 24 hours
Period: Overall Study
Arm/Group | GW-1000-02
Started | 137
Completed | 70
Not Completed | 67
Not completed — Lack of Efficacy | 26
Not completed — Adverse Event | 18
Not completed — Moved out of area | 6
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 4
Not completed — Symptom control without study medication | 2
Not completed — Unable to make journey | 1
Not completed — Death | 1
Not completed — Cannabis affecting job | 1
Not completed — Felt more alter without study medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | GW-1000-02
Number analyzed (Participants) | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 127
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.69 (9.531)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 54
Region of Enrollment [Number; unit: participants]
  United Kingdom | 137

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events as a Measure of Patient Safety
Description: The number of patients who experienced an adverse event during the course of this extension study is presented
Time Frame: up to1206 days
Population: All subjects who took at least one dose of study medication after the end of the Part B open-label phase of the acute study, and yielded on-treatment efficacy data was classed as the efficacy and safety population.
Measure: Number; unit: participants
Groups:
- GW-1000-02: Contains THC (27 mg/ml) and CBD (25 mg/ml). Subjects received study medication delivered in 100 μl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three hour period and 48 actuations (THC 130 mg:CBD 120 mg) in 24 hours
Arm/Group | GW-1000-02
Number analyzed (Participants) | 137
participants | 126

2. Secondary Outcome: Mean Number of Sprays of Study Medication Taken During the Last 6 Days of Treatment
Description: A categorical summary was produced of the mean number of sprays per day during the last six days of treatment, and the mean number of sprays was rounded to the nearest whole number for categorisation.
Time Frame: up to 1206 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sprays of study medication
Arm/Group | GW-1000-02
Number analyzed (Participants) | 137
sprays of study medication | 8.09 (7.91)

3. Secondary Outcome: Change From Baseline in Mean Intoxication 100 mm Visual Analogue Scale Scores at Week 18.
Description: Intoxication levels were recorded on a Visual Analogue Scale, where 0 equals 'no intoxication' and 10 equals 'extreme intoxication'. A decrease in score indicates an improvement in intoxication levels.
Time Frame: 18 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 121
units on a scale | 2.65 (14.15)

4. Secondary Outcome: Investigator Assessed Global Severity Score at Week 18
Description: The investigator rated the global severity of the subject's primary condition since entry into the study using a five-point verbal rating scale-5: 1=much worse, 2=worse, 3=no change, 4=better, 5=much better. The number of patients which were considered better or much better (scores 4 and 5) at week 18 of the study better is presented.
Time Frame: week 18
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 135
participants | 92

5. Secondary Outcome: Change From Baseline in the Mean Pain 100 mm Visual Analogue Scale Score at Week 18
Description: A clinical assessment of pain was made at each study visit using a 100 mm Visual Analogue Scale, where 0 = no pain and 100 = worst possible pain. A decrease in score indicates an improvement.
Time Frame: week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 74
units on a scale | -31.34 (27.20)

6. Secondary Outcome: Change From Baseline in the Mean Spasticity 100 mm Visual Analogue Scale Score at Week 18
Description: A clinical assessment of spasticity was made at each study visit using a 100 mm Visual Analogue Scale, where 0 = no spasticity and 100 = worst possible spasticity. A decrease in score indicates an improvement.
Time Frame: week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 118
units on a scale | -27.81 (24.46)

7. Secondary Outcome: Change From Baseline in the Mean Tremor 100 mm Visual Analogue Scale Score at Week 18
Description: A clinical assessment of tremor was made at each study visit using a 100 mm Visual Analogue Scale, where 0 = no tremor and 100 = worst possible tremor. A decrease in score indicates an improvement.
Time Frame: week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 43
units on a scale | -26.23 (23.90)

8. Secondary Outcome: Change From Baseline in the Mean Bladder Problems 100 mm Visual Analogue Scale Score at Week 18
Description: A clinical assessment of bladder problems was made at each study visit using a 100 mm Visual Analogue Scale, where 0 = no bladder problems and 100 = worst possible bladder problems. A decrease in score indicates an improvement.
Time Frame: 18 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 96
units on a scale | -33.60 (25.12)

ADVERSE EVENTS:
Time Frame: All adverse events occurring from during the extension study (up to 1049 days) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | GW-1000-02
Serious Adverse Events (participants affected / at risk) | 23/137
Other Adverse Events (participants affected / at risk) | 127/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=137)
Urinary Tract Infection Not Otherwise Specified (NOS) (Infections and infestations) | 4
Pneumonia NOS (Infections and infestations) | 1
Bone infection NOS (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 3
Balance Impaired NOS (Nervous system disorders) | 2
Convulsions NOS (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Fall (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Weakness (General disorders) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Lower Limb Fracture NOS (Injury, poisoning and procedural complications) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Muscle Weakness NOS (Musculoskeletal and connective tissue disorders) | 2
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Cancer Stage Unspecified (excl metastatic tumours to lung) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vomiting NOS (Gastrointestinal disorders) | 2
Diarrhoea NOS (Gastrointestinal disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Biliary Cirrhosis Primary (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Panic Attack (Psychiatric disorders) | 1
Psychotic Disorder NOS (Psychiatric disorders) | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2
Deep Vein Thrombosis NOS (Vascular disorders) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.6% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=137)
ORAL PAIN (Gastrointestinal disorders) | 32
DIARRHOEA NOS (Gastrointestinal disorders) | 27
NAUSEA (Gastrointestinal disorders) | 24
VOMITING NOS (Gastrointestinal disorders) | 16
GLOSSODYNIA (Gastrointestinal disorders) | 15
ORAL MUCOSAL DISORDER (Gastrointestinal disorders) | 15
CONSTIPATION (Gastrointestinal disorders) | 12
DRY MOUTH (Gastrointestinal disorders) | 11
ORAL DISCOMFORT (Gastrointestinal disorders) | 9
MOUTH ULCERATION (Gastrointestinal disorders) | 8
DYSPEPSIA (Gastrointestinal disorders) | 7
LOOSE STOOLS (Gastrointestinal disorders) | 7
TOOTHACHE (Gastrointestinal disorders) | 7
TOOTH DISCOLOURATION (Gastrointestinal disorders) | 6
FALL (General disorders) | 21
FATIGUE (General disorders) | 16
WEAKNESS (General disorders) | 11
LETHARGY (General disorders) | 10
APPLICATION SITE IRRITATION (General disorders) | 9
APPLICATION SITE PAIN (General disorders) | 6
MALAISE (General disorders) | 6
FEELING ABNORMAL (General disorders) | 5
URINARY TRACT INFECTION NOS (Infections and infestations) | 56
NASOPHARYNGITIS (Infections and infestations) | 37
LOWER RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 13
TOOTH CARIES NOS (Infections and infestations) | 9
BACTERIAL INFECTION NOS (Infections and infestations) | 8
BLADDER INFECTION NOS (Infections and infestations) | 6
VAGINAL CANDIDIASIS (Infections and infestations) | 6
VIRAL INFECTION NOS (Infections and infestations) | 5
WEIGHT DECREASED (Investigations) | 13
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 10
ANOREXIA (Metabolism and nutrition disorders) | 7
PAIN IN LIMB (Musculoskeletal and connective tissue disorders) | 17
MUSCLE WEAKNESS NOS (Musculoskeletal and connective tissue disorders) | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 5
PERIPHERAL SWELLING (Musculoskeletal and connective tissue disorders) | 5
DIZZINESS (Nervous system disorders) | 30
HEADACHE NOS (Nervous system disorders) | 23
BALANCE IMPAIRED NOS (Nervous system disorders) | 21
MULTIPLE SCLEROSIS AGGRAVATED (Nervous system disorders) | 16
DYSGEUSIA (Nervous system disorders) | 13
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 12
DISTURBANCE IN ATTENTION (Nervous system disorders) | 9
SOMNOLENCE (Nervous system disorders) | 9
SYNCOPE (Nervous system disorders) | 9
MEMORY IMPAIRMENT (Nervous system disorders) | 6
SHORT-TERM MEMORY LOSS (Psychiatric disorders) | 9
DEPRESSED MOOD (Psychiatric disorders) | 7
DISORIENTATION (Psychiatric disorders) | 6
INSOMNIA (Psychiatric disorders) | 5
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 8
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 5
CONTUSION (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.